CLINICAL TRIAL: NCT00304395
Title: Pulmonary Infections Masquerading as Community-Acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Daniel M. Musher MD, Principal Investigator, Michael E. DeBakey VA Medical Center
Other Study IDs: H-17555
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia
Keywords: Community Acquired Pneumonia; CAP
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to identify cases from patients who have been referred for consultation to the Infectious Disease Section at the VAMC, Houston, and to compare them with other cases of CAP in order to determine whether there are features that might enable non-CAP cases to be distinguished from CAP.

DETAILED DESCRIPTION:
Guidelines to treat community acquired pneumonia (CAP) have been developed and widely promulgated by important professional societies in the past 10 years. The impetus to do so came from the observation that practicing physicians were using a wide array of approaches to this common infection, many of which were substandard.

The Infectious Disease Society of America (IDSA) and American Thoracic Society (ATS) have been leaders in this field, publishing recommendations separately between 1993 and 2003. The PI served on the IDSA committee and coauthored the publication in 2000 and the update in 2003. In 2004, a decision was made by the two professional societies to merge the committees and make a single joint set of recommendations; the PI is a member of that joint committee and a new document is being prepared for publication.

The PI has observed a tendency to apply these guidelines to cases that might masquerade as CAP but are actually attributable to other conditions, such as lung cancer, tuberculosis and histoplasmosis. Further, the recommendations do not adequately cover pneumonia due to Staphylococcus aureus.

The purpose of the research is to identify cases from the consult records of the Infectious Disease Section at the VAMC, Houston, and to compare them with other cases of CAP in order to determine whether there are features that might enable non-CAP cases to be distinguished from CAP.

ELIGIBILITY:
Inclusion Criteria:

* subjects who were seen in calendar year 2004 because they were thought to have CAP, but who, upon further evaluation, plainly did not, and consultation was sought.
* case control is diagnosis of CAP with verification by all or nearly all of the following features: presence of cough, increased sputum, fever, leukocytosis and a distinct new pulmonary infiltrate.

Exclusion Criteria:

* among the case controls, if the diagnosis of CAP was made despite the absence of the cardinal features of CAP, as cited above, the investigators will not include the case.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Pulmonary infections.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2004-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, M.D., Principal Investigator — Baylor College of Medicine, Houston VA Medical Center
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States